CLINICAL TRIAL: NCT02641639
Title: FOCUS: A Multicenter, Multinational, Double-Blind, 2-Arm, Randomized, Phase 2/3, Study of Physician's Choice Chemotherapy ([PCC] Weekly Paclitaxel or Pegylated Liposomal Doxorubicin [PLD]) Plus Bevacizumab and CA4P Versus PCC Plus Bevacizumab and Placebo for Subjects With Platinum-Resistant, Recurrent Epithelial Ovarian, Primary Peritoneal or Fallopian Tube Cancer
Brief Title: FOCUS: PCC + Bevacizumab + CA4P Versus PCC + Bevacizumab + Placebo for Subjects With Platinum Resistant Ovarian Cancer
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: The study was terminated early due to the lack of efficacy and the study sponsor's decision to no longer continue the study
Sponsor: Mateon Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: OX4325
Record Dates: First submitted 2015-12-21; First posted 2015-12-29 (Estimated); Results first posted 2025-03-24 (Actual); Last update posted 2025-03-24 (Actual); Status verified 2025-03

CONDITIONS: Platinum Resistant Ovarian Cancer
MeSH Terms: interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Fosbretabulin tromethamine (Active Comparator): Physician's choice chemotherapy (weekly Paclitaxel or Pegylated Liposomal Doxorubicin [PLD]) plus bevacizumab and CA4P
  Interventions: Drug: Fosbretabulin tromethamine
- Placebo (Placebo Comparator): Physician's choice chemotherapy (weekly Paclitaxel or Pegylated Liposomal Doxorubicin [PLD]) plus bevacizumab and placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Fosbretabulin tromethamine — CA4P is a synthetic phosphorylated prodrug of CA4, a naturally occurring derivative of the South African willow tree, combretum caffrum. CA4P targets pre-existing tumor vasculature, resulting in an acute, reversible reduction in TBF that leads to central necrosis within tumors.
  Other Names: Fosbretabulin Combretastatin A4-Phosphate, CA4P
  Arms: Fosbretabulin tromethamine
Drug: Placebo — Saline for infusion
  Other Names: Saline for infusion
  Arms: Placebo

SUMMARY:
This is a multicenter, multinational, randomized, double-blind, 2-arm, parallel-group, Phase 2/3 study to evaluate the efficacy and safety of PCC plus bevacizumab and CA4P versus PCC plus bevacizumab and placebo in subjects with platinum-resistant ovarian cancers (prOC). Subjects with platinum-resistant, recurrent, epithelial ovarian, primary peritoneal or fallopian tube cancer will be randomized 1:1 to receive PCC plus bevacizumab and CA4P or PCC plus bevacizumab and placebo. Subjects will be stratified by selected chemotherapy (PLD vs. paclitaxel), platinum free interval (< 3 vs. 3 to 6 months from last platinum therapy to subsequent progression), and line of therapy (2nd vs. 3rd). This is a 2-part study, consisting of a Phase 2, exploratory study (Part 1) followed by a Phase 3, pivotal study (Part 2). Both parts of the study will have similar overall design. Approximately 80 subjects will be randomized into Part 1 and approximately 356 subjects will be randomized into Part 2.

DETAILED DESCRIPTION:
This is a multicenter, multinational, randomized, double-blind, 2-arm, parallel-group, Phase 2/3 study to evaluate the efficacy and safety of PCC plus bevacizumab and CA4P versus PCC plus bevacizumab and placebo in subjects with platinum-resistant ovarian cancers (prOC). Subjects with platinum-resistant, recurrent, epithelial ovarian, primary peritoneal or fallopian tube cancer will be randomized 1:1 to receive PCC plus bevacizumab and CA4P or PCC plus bevacizumab and placebo. Subjects will be stratified by selected chemotherapy (PLD vs. paclitaxel), platinum free interval (< 3 vs. 3 to 6 months from last platinum therapy to subsequent progression), and line of therapy (2nd vs. 3rd). This is a 2-part study, consisting of a Phase 2, exploratory study (Part 1) followed by a Phase 3, pivotal study (Part 2). Both parts of the study will have similar overall design. Approximately 80 subjects will be randomized into Part 1 and approximately 356 subjects will be randomized into Part 2.

All subjects randomized will receive bevacizumab 10 mg/kg intravenously (IV) on Days 1 and 15, repeated every 4 weeks (q4wk) and PCC with paclitaxel 80 mg/m2 IV on Days 1, 8, 15 and 22, repeated q4wk, or paclitaxel 80 mg/m2 IV on Days 1, 8, 15, repeated q4wk or PLD 40 mg/m2 IV on Day 1, repeated q4wk. Subjects in the Treatment Arm will also receive CA4P 60 mg/m2 on the same day as bevacizumab (Days 1 and 15, repeated q4wk), while subjects in the Control Arm will receive placebo on those days.

Order of dosing will follow the guidance listed below during this study when bevacizumab and CA4P / Placebo are dosed the same day as PCC,

* Bevacizumab followed by CA4P / Placebo followed after 1-3 hours by paclitaxel,
* PLD followed by bevacizumab followed by CA4P / Placebo Subjects will continue randomized treatment until disease progression, unacceptable toxicity, investigator decision, withdrawal of consent, or sponsor discontinues study for any reason. Subjects will undergo tumor assessments (RECIST) at baseline and every 8 weeks and CA-125 levels at baseline and every 4 weeks.

The primary endpoint is PFS. Secondary endpoints include ORR, OS, proportion of subjects who remain progression free at 6, 9, and 12 months, and safety. Endpoints will be compared between the Treatment Arm and the Control arm. The study duration is estimated to last approximately 3 years.

This study will have 2 parts with the same overall design. Part 1 will enroll up to approximately 80 subjects and will include multiple interim analyses to test the safety and efficacy assumptions in this specific subject population. Upon meeting certain efficacy criteria in Part 1, the protocol will be amended and additional sites added in order to enroll an additional 356 subjects into Part 2 of the study. Subjects enrolled in Part 2 will be analyzed separately and used as a stand-alone confirmatory efficacy study.

ELIGIBILITY:
Inclusion:

1. Signed informed consent form (ICF)
2. Age ≥ 18 years (Age ≥ 19 years if required by local regulatory authorities)
3. ECOG PS of 0-1
4. Histologically or cytologically-confirmed epithelial ovarian, fallopian tube or primary peritoneal cancer in recurrent stage
5. prOC (platinum-resistant ovarian cancers) defined as progression within > 1 to < 6 months (+ 2 weeks) of completing previous cycle of primary platinum-based therapy, or during or within < 6 months (+ 2 weeks) of starting additional platinum based therapies
6. Received ≥ 1 but ≤ 3 prior platinum-based regimens
7. Measurable disease according to RECIST 1.1
8. Left ventricular ejection fraction (LVEF) greater than or equal to at least 45% at baseline assessment if subject is receiving PLD, and/or anthracycline is a concomitant medication
9. No evidence of active (progressing) brain metastasis. (Treated brain metastasis allowed with a posttreatment magnetic resonance imaging (MRI) or Computed Tomography (CT) of brain showing no active (progressing) brain metastasis). Treatment of brain metastasis may include surgery, radiosurgery (linear accelerator (LINAC), gamma knife), or whole brain irradiation. Surgery for brain metastasis must be > 8 weeks from study entry
10. Hemoglobin > 9 g/dl. Erythroid growth factors should not have been used in the 2 weeks prior to study entry. Red blood cell transfusions are permitted to maintain the hemoglobin level > 9 g/dl
11. Adequate bone marrow function in the investigator's opinion
12. Adequate hepatic function defined by the following:

    * Total bilirubin < 2 x Upper Limit of Normal (ULN)
    * Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) < 2.5 X ULN for the referenced lab (< 5 X ULN for subjects with liver metastases)
13. Adequate renal function defined by the following:

    - Serum creatinine < 2 X ULN for the referenced lab
14. Subjects of childbearing potential must have a negative serum pregnancy test prior to study entry and must be practicing a highly effective form of contraception
15. At least 2 weeks since prior radiotherapy and has recovered from any Grade 3 toxicities
16. Life expectancy ≥ 12 weeks

Exclusion:

1. Subjects who have received prior CA4P therapy
2. Previously having failed treatment with bevacizumab combined with the intended PCC.

   - For clarity: Investigators should not select a bevacizumab + PCC combination for the FOCUS trial if the patient has previously failed that same regimen, however they may select a new PCC regimen to combine with bevacizumab. For example, a patient who failed bevacizumab + weekly paclitaxel would be allowed to enroll in FOCUS only if they are assigned to bevacizumab + PLD for the study.
3. Previous treatment with greater than three traditional chemotherapy treatment regimens
4. Untreated brain metastasis or leptomeningeal brain metastasis
5. Solid organ or bone marrow transplant
6. Primary platinum-refractory disease (defined as progression during dosing or within one (1) month of completing the last cycle of patients first platinum-containing regimen)
7. > Grade 2 peripheral neuropathy
8. Current thrombotic or hemorrhagic disorder/event or history of prior event within 6 months of start of Screening
9. History of prior cerebrovascular event, (including transient ischemic attack) within 6 months of start of Screening
10. Recent history (within 6 months of start of Screening) of angina pectoris, myocardial infarction (including non-Q wave MI), or NYHA Class III and IV congestive heart failure
11. History of torsade de pointes, ventricular tachycardia or fibrillation, pathologic sinus bradycardia (<60 bpm), heart block (excluding 1st degree block, benign PR interval prolongation only), congenital long QT syndrome or new ST segment elevation or depression or new Q wave on ECG
12. Known uncontrolled HIV infection
13. Uncontrolled, clinically significant active infection
14. Serious non-healing wound, ulcer or bone fracture
15. Subjects with known hypersensitivity to any of the components of CA4P, paclitaxel, PLD, or bevacizumab (paclitaxel and PLD dependent on whether PI plans they will be dosed with that PCC)
16. Subjects who are currently or planning on receiving concurrent investigational therapy or who have received investigational therapy for any indication within 30 days of the first scheduled day of dosing
17. Subjects with any other intercurrent medical condition, including mental illness or substance abuse, deemed by the Investigator to be likely to interfere with a subject's ability to provide informed consent, cooperate and participate in the study, or to interfere with the interpretation of the study results
18. Subjects with other invasive malignancies, with the exception of non-melanoma skin cancer, or with previous cancer treatment that contraindicates this protocol therapy within last 3 years
19. Prior radiation therapy to the pelvis or abdomen within 4 weeks of entry into the study
20. History of fistula, gastrointestinal (GI) perforation or intra-abdominal abscess, or invasive disease/metastases of the bowel which in the investigators opinion may increase the risk of GI perforation with bevacizumab treatment.
21. Uncontrolled hypertension (HTN)

    - Sustained BP greater than 150 mmHG SBP / 100 mmHG DBP
22. Uncontrolled elevated proteinuria levels in the investigator's opinion
23. Corrected QT interval ([QTc] Fridericia) > 480 ms
24. Significant vascular disease or recent peripheral arterial thrombosis
25. Subjects with active bleeding or pathologic conditions that carry high risk of bleeding
26. Subjects who are pregnant or lactating

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2017-10 (Actual); Study Completion 2017-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Harish Dave, MD, Study Director — Medical Monitor
Locations (40):
- United States (36):
  - University of Alabama at Birmingham Comprehensive Cancer Center, Birmingham, Alabama
  - Mitchell Cancer Institute - USA Health System, Mobile, Alabama
  - Arizona Oncology Associates, PC - HAL, Phoenix, Arizona
  - Arizona Oncology Associates, PC - HOPE, Tucson, Arizona
  - University of Arizona Cancer Center, Tucson, Arizona
  - Oncology Institute of Hope and Innovation, Lynwood, California
  - University of California Irvine, Orange, California
  - California Pacific Medical Center, Research Institute, San Francisco, California
  - Sansum Clinic, Santa Barbara, California
  - Rocky Mountain Cancer Centers, LLP, Lakewood, Colorado
  - Hartford Health Care Cancer Institute; Affiliate Memorial Sloan Kettering, Hartford, Connecticut
  - Stamford Hospital - Bennett Cancer Center, Stamford, Connecticut
  - Sylvester Comprehensive Cancer Center University of Miami, Miami, Florida
  - Baptist Health Medical Group Oncology, LLC, Miami, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - Augusta University, Augusta, Georgia
  - Maine Medical Center, Scarborough, Maine
  - Mercy Medical Center; The Institute for Cancer Care, Baltimore, Maryland
  - HCA Midwest Division - Sarah Cannon Cancer Institute, Kansas City, Missouri
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Gabrail Cancer Center, Canton, Ohio
  - Oklahoma Heath Sciences Center - Stephenson Cancer Center, Oklahoma City, Oklahoma
  - Tulsa Cancer Institute, Tulsa, Oklahoma
  - OHSU Center for Women's Health & Knight Cancer Institute, Portland, Oregon
  - Willamette Valley Cancer Institute, Springfield, Oregon
  - Lehigh Valley Hospital, John and Dorothy Morgan Cancer Center; Affiliate Memorial Sloan Kettering, Allentown, Pennsylvania
  - The Western Pennsylvania Hospital, Pittsburgh, Pennsylvania
  - Gibbs Cancer Center & Research Institute Spartanburg Medical Center, Spartanburg, South Carolina
  - Texas Oncology, P.A., Austin, Texas
  - Texas Oncology, Bedford, Texas
  - Dallas County Hospital District d/b/a Parkland Health and Hospital System, Dallas, Texas
  - Simmons Comprehensive Cancer Center; UT Southwestern Medical Center, Dallas, Texas
  - Texas Oncology, P.A., Dallas, Texas
  - Texas Oncology San Antonio, San Antonio, Texas
  - Texas Oncology, P.A., The Woodlands, Texas
  - Texas Oncology, P.A., Tyler, Texas
- UZ Leuven, Leuven, Belgium
- Germany (3):
  - Universitätsklinikum Erlangen, Erlangen
  - Universitätsklinikum Essen (AöR) Klinik für Frauenheilkunde und Geburtshilfe, Essen
  - Universitäts-Frauenklinik Dept. für Frauengesundheit, Tübingen

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Fosbretabulin Tromethamine | Placebo
Started | 34 | 36
Completed | 34 | 36
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Fosbretabulin Tromethamine | Placebo | Total
Number analyzed (Participants) | 34 | 36 | 70
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 14 | 17 | 31
  >=65 years | 20 | 19 | 39
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.9 (8.02) | 63.2 (8.05) | 65 (8.18)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34 | 36 | 70
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 5 | 7
  Not Hispanic or Latino | 32 | 31 | 63
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 3 | 7
  White | 30 | 32 | 62
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Baseline Tumor Diameter Sum (cm) [Mean (Standard Deviation); unit: cm] | 80.1 (64.17) | 67.5 (40.90) | 73.7 (53.44)

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival
Description: The primary efficacy parameter in this study is statistically meaningful PFS, defined as the time from the date of randomization until patient discontinuation or death from any cause.
Time Frame: 12 Months
Measure: Mean (Full Range); unit: days
Arm/Group | Fosbretabulin Tromethamine | Placebo
Number analyzed (Participants) | 34 | 36
days | 116.9 [19 to 292] | 120.4 [19 to 239]

2. Secondary Outcome: Improvement in Objective Response Rate
Description: Improvement in objective response rate (ORR). The ORR will be defined as the proportion of subjects with a confirmed complete response (CR) or confirmed partial response (PR) per RECIST 1.1 criteria, based upon the best response. The ORR will be determined based on investigator assessment according to RECIST 1.1 criteria and/or GCIG CA-125 criteria.
Time Frame: 12 Months
Measure: Count of Participants; unit: Participants
Arm/Group | Fosbretabulin Tromethamine | Placebo
Number analyzed (Participants) | 34 | 36
Participants | 8 | 13

3. Secondary Outcome: Overall Survival (OS)
Description: Evaluation of overall survival (OS)
Time Frame: 12 Months
Measure: Count of Participants; unit: Participants
Arm/Group | Fosbretabulin Tromethamine | Placebo
Number analyzed (Participants) | 34 | 36
Participants
  Dies while on study | 6 | 4
  Censored | 28 | 32

4. Secondary Outcome: Proportion of Subjects Who Remain Progression-free at 12 Months
Description: Assessment of the proportion of subjects who remain progression-free at 12 months on the regimen of PCC plus bevacizumab and CA4P compared with PCC plus bevacizumab and placebo
Time Frame: 12 Months
Measure: Count of Participants; unit: Participants
Arm/Group | Fosbretabulin Tromethamine | Placebo
Number analyzed (Participants) | 34 | 36
Participants | 22 | 24

5. Secondary Outcome: Incidence of Treatment-Emergent Adverse Events (Safety and Tolerability) of PCC Plus Bevacizumab and CA4P Versus PCC Plus Bevacizumab and Placebo
Description: To evaluate the Incidence of Treatment-Emergent Adverse Events of PCC plus bevacizumab and CA4P versus PCC plus bevacizumab and placebo as measured by aggregate reporting of the number of patient with abnormal findings on (physical exams, vital signs, laboratory measures, ECG, Eastern Cooperative Oncology Group (ECOG) performance status (PS)) and/or analysis of the incidence of adverse events (AEs) using the National Cancer Institute (NCI)-Common Terminology Criteria for AEs (CTCAE) version 4.03.
Time Frame: 12 Months
Measure: Count of Participants; unit: Participants
Arm/Group | Fosbretabulin Tromethamine | Placebo
Number analyzed (Participants) | 34 | 36
Participants | 28 | 30

ADVERSE EVENTS:
Time Frame: 1 year, 3 months
Description: MedDRA System Organ Class
Arm/Group | Fosbretabulin Tromethamine | Placebo
All-Cause Mortality (participants affected / at risk) | 6/34 | 4/36
Serious Adverse Events (participants affected / at risk) | 10/34 | 11/36
Other Adverse Events (participants affected / at risk) | 28/34 | 30/36
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Fosbretabulin Tromethamine (N=34) | Placebo (N=36)
Cardiac disorders (Cardiac disorders) | 1 | 1
Gastrointestinal disorders (Eye disorders) | 3 | 3
Infections and infestations (Infections and infestations) | 3 | 5
Metabolism and nutrition disorders (Metabolism and nutrition disorders) | 3 | 1
Psychiatric disorders (Psychiatric disorders) | 2 | 0
Respiratory, thoracic and mediastinal disorders (Respiratory, thoracic and mediastinal disorders) | 3 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Fosbretabulin Tromethamine (N=34) | Placebo (N=36)
Anemia (Blood and lymphatic system disorders) | 4 | 4
Constipation (Gastrointestinal disorders) | 6 | 4
Diarrhea (Gastrointestinal disorders) | 4 | 7
Nausea (Gastrointestinal disorders) | 11 | 7
Stomatitis (Gastrointestinal disorders) | 5 | 5
Fatigue (General disorders) | 11 | 10
Edema peripheral (General disorders) | 4 | 6
Hypomagnesemia (Metabolism and nutrition disorders) | 2 | 4
Headache (Nervous system disorders) | 7 | 9
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 | 5
Erythema (Skin and subcutaneous tissue disorders) | 1 | 4
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 5 | 9
Hot flush (Vascular disorders) | 3 | 4
Hypertension (Vascular disorders) | 13 | 12

LIMITATIONS AND CAVEATS:
Early termination leading to small numbers of subjects analyzed

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-03-21): https://cdn.clinicaltrials.gov/large-docs/39/NCT02641639/Prot_SAP_000.pdf